CLINICAL TRIAL: NCT05147649
Title: Functional Magnetic Resonance Imaging in Patients With Obstructive Sleep Apnea Syndrome, With and Without CPAP, During Wakefulness - Impact on Cognitive Functions
Brief Title: Functional Magnetic Resonance Imaging in Patients With Obstructive Sleep Apnea Syndrome
Acronym: IRM SAOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PA21141*
Record Dates: First submitted 2021-11-29; First posted 2021-12-07 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-OSAS patients (Active Comparator): Patients without OSAS (Apnea-Hypopnea Index (AHI) < 15/h and absence of excessive daytime sleepiness with Epworth score <11)
  Interventions: Diagnostic Test: functional magnetic resonance imaging
- OSAS patients (Experimental): Patients with severe OSAS with an Apnea-Hypopnea Index (AHI) > 30/h
  Interventions: Diagnostic Test: functional magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: functional magnetic resonance imaging — functional magnetic resonance imaging

SUMMARY:
The obstructive sleep apnea syndrome (OSAS) involves recurrent sleep-related upper airways (UA) collapse. UA mechanical properties and neural control are altered, imposing a mechanical load on inspiration. UA collapse does not occur during wakefulness, hence arousal-dependent compensation. Experimental inspiratory loading in normal subjects elicits respiratory-related cortical activity during wakefulness. The objective of this study is to test whether awake OSAS patients would exhibit a similar cortical activity. Whether or not such cortical compensatory mechanisms have cognitive consequences would be also analyze.

ELIGIBILITY:
Inclusion criteria :

1. OSAS patients

   * severe OSAS with an Apnea-Hypopnea Index (AHI) > 30/h
   * without CPAP treatment
2. Non-OSAS patients

   * absence of OSAS (AHI < 15/h and absence of excessive daytime sleepiness with Epworth score <11)

Non-inclusion criteria :

* < 18 years old
* >75 years old
* left-handed
* BMI> 40 kg/m²
* another sleep disorder
* central component of sleep apnea syndrome (central apnea index> 5 / h)
* current or past neurological pathology
* respiratory pathology (obstructive ventilatory disorder, restrictive ventilatory disorder, hypercapnia)
* MRI contraindication (metallic foreign body, claustrophobia, pregnant woman, etc.)
* taking drugs that can modify the BOLD signal on MRI (psychotropic drugs, vasodilators, vasoconstrictors, etc.),
* uncorrected sensory impairment (vision or hearing)
* protected by law.

Exclusion criteria :

* pregnant woman according to the positive beta-hCG test result
* left-handed following the laterality questionnaire
* MINI results showing:

  * a current mood episode
  * a current disorder of the use of psychoactive substances or in the last 6 months (excluding tobacco)
  * an eating disorder
  * a diagnosis of bipolar disorder, current or past schizophrenia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-07-02 (Estimated)

PRIMARY OUTCOMES:
Premotor cortex activation in OSAS patients without CPAP | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided